CLINICAL TRIAL: NCT02624700
Title: Phase 2 Study of Pemetrexed and Sorafenib for Treatment of Recurrent or Metastatic Triple Negative Breast Cancer
Brief Title: 2nd Line Treatment With Pemetrexed and Sorafenib for Recurrent or Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eli Lilly and Company (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14-10790; HM20005967; NCI-2015-02190 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: ER-negative; PgR-negative; Human epidermal growth factor receptor 2 (HER2-negative); Triple Negative Breast Cancer; HER2-negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Pemetrexed; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Pemetrexed + Sorafenib (Experimental): Pemetrexed 500 mg/m2 IV Day 1 + Sorafenib 400mg PO twice each day on Days 1-5 of each 14-day cycle
  Interventions: Drug: Experimental Arm A: Pemetrexed; Drug: Experimental Arm A: Sorafenib
- B: Pemetrexed + Sorafenib (Experimental): Pemetrexed 375mg/m2 intravenously (IV) Day 1 + Sorafenib 200mg by mouth twice daily on days 1-5, every 21 days of each cycle.
  Interventions: Drug: Experimental Arm B: Pemetrexed; Drug: Experimental Arm B: Sorafenib

INTERVENTIONS:
Drug: Experimental Arm A: Pemetrexed — Treatment schedule is administered on day 1 of each 14-day cycle by Intravenous infusion over 10 minutes with a dose of 500 mg/m2. If necessary, the duration of the pemetrexed infusion may be extended to a maximum of 20 minutes.
  Other Names: Alimta
  Arms: A: Pemetrexed + Sorafenib
Drug: Experimental Arm A: Sorafenib — Treatment schedule is administered twice daily by mouth on an empty stomach on days 1-5 of each 14-day cycle with a dose of 400 mg.
  Other Names: Nexavar
  Arms: A: Pemetrexed + Sorafenib
Drug: Experimental Arm B: Pemetrexed — Treatment schedule is administered on day 1 of each 21-day cycle by Intravenous infusion over 10 minutes with a dose of 375 mg/m2. If necessary, the duration of the pemetrexed infusion may be extended to a maximum of 20 minutes.
  Other Names: Alimta
  Arms: B: Pemetrexed + Sorafenib
Drug: Experimental Arm B: Sorafenib — Treatment schedule is administered twice daily by mouth on an empty stomach on days 1-5 of each 21-day cycle with a dose of 200 mg.
  Other Names: Nexavar
  Arms: B: Pemetrexed + Sorafenib

SUMMARY:
This phase 2 clinical trial will evaluate the efficacy of the combination of pemetrexed and sorafenib in patients with recurrent or metastatic Triple Negative Breast Cancer (TNBC). Candidate pharmacodynamic and predictive biomarkers will also be evaluated.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, phase 2 study of a regimen of dose-dense pemetrexed and sorafenib to determine the objective response rate in patients with recurrent or metastatic TNBC. Eligible patients will be those who have had disease progression during or after treatment for recurrent or metastatic disease with one previous cytotoxic chemotherapy regimen. Additionally, patients with disease progression or recurrence during or within 6 months of completion of adjuvant or neoadjuvant therapy are also eligible. Correlative studies will be conducted using blood samples and archived tumor samples.

Simon's two-stage design will be utilized in this study. In the first stage, if there are ≤ 3 patients of the first 18 efficacy-evaluable patients who have a partial or complete response, then the trial will end for futility. If ≥ 4 patients have a partial or complete response, patient accrual will continue in the second stage to add 10 more efficacy-evaluable patients.

The total sample size for the Simon's two-stage design is 35 patients. Based on enrollment of 2-3 patients per month, the expected enrollment period will be about 12-18 months.

Patients were enrolled in 2 sequential groups, referred to as "arms" for the purposes of reporting results by group. The initial group of patients were enrolled in what is referred to here as Arm A. After a study amendment patients were enrolled in what is referred to here as Arm B.

ELIGIBILITY:
Inclusion Criteria

* Unresectable adenocarcinoma of the breast involving chest wall, regional nodes, or distant site
* Breast cancer determined to be estrogen receptor (ER)-negative and progesterone receptor (PgR)-negative defined for this study as < 10% tumor staining by immunohistochemistry (IHC) (Note: Eligibility should be based on the ER and PgR status reported at the time of the most recent biopsy or resection).
* Breast cancer determined to be HER2-negative per current American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) HER2 Guidelines (Note: Eligibility should be based on the HER2 status reported at the time of the most recent biopsy or resection).
* At least one prior regimen for treatment of recurrent or metastatic disease (Note: Prior regimen for recurrent or metastatic disease is not required if the patient had disease progression or recurrence during or within the first 6 months following completion of adjuvant or neoadjuvant chemotherapy.)
* Measurable disease per RECIST v1.1
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Ability to swallow oral medications
* Adequate bone marrow function as defined below:
* Absolute neutrophil count (ANC) ≥ 1,200/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 9.0 g/dL, which must be stable in the opinion of the investigator without a history of transfusion dependence.
* Adequate renal function as defined below:
* Calculated creatinine clearance ≥ 45 mL/min
* Adequate hepatic function as defined below:
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the laboratory
* Aspartate aminotransferase (AST) ≤ 3 x ULN for the laboratory, except in the presence of known hepatic metastasis, wherein the AST may be ≤ 5 x ULN
* Alanine aminotransferase (ALT) ≤ 3 x ULN for the laboratory, except in the presence of known hepatic metastasis, wherein the ALT may be ≤ 5 x ULN
* Serum B12 and folate levels ≥ lower limit of normal (LLN) for the laboratory (Note: Patients may begin B12 and folic acid supplementation and be reconsidered for participation in the study when levels are ≥ LLN for the laboratory).
* Ability to take folic acid, vitamin B12, and dexamethasone according to the protocol instructions
* Ability to interrupt chronic non-steroidal anti-inflammatory drugs (NSAIDs) beginning 2 days before (5 days before for long-acting NSAIDs) and continuing for 2 days following administration of each pemetrexed dose
* Toxicities from previous cancer therapies resolved to ≤ grade 1 unless specified otherwise in the inclusion or exclusion criteria
* Women who are not postmenopausal or have not undergone hysterectomy must have a documented negative serum pregnancy test within 7 days prior to initiating study treatment. Note: Postmenopausal is defined as one or more of the following:
* Age ≥ 60 years
* Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
* Bilateral oophorectomy
* A woman of child-bearing potential (WCBP) and a male patient with partner who is a WCBP must agree to use a medically accepted method for preventing pregnancy for the duration of study treatment and for 2 months following completion of study treatment.
* Ability to understand and willingness to sign the consent form written in English

Exclusion Criteria

* Any investigational agent within 4 weeks prior to initiating study treatment
* Anticancer therapy within 2 weeks prior to initiating study treatment
* Plans for concurrent anticancer therapy except as permitted in Section 6.7.11
* Known or presumed intolerance of pemetrexed or sorafenib
* Known or suspected malabsorption condition or obstruction
* Brain metastases meeting either of the following exclusion criteria:
* Untreated brain metastases
* After completion of brain-directed therapy, the patient has not been able to tolerate discontinuation of steroids or a decrease in steroid dose
* Leptomeningeal metastasis
* Any documented history of clinically identifiable thrombotic, embolic, venous, or arterial events such as cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or pulmonary embolism within 6 months prior to initiating study treatment (Note: Patients with an asymptomatic catheter-related thrombus or a tumor-associated thrombus of locally-involved vessels or with incidental asymptomatic filling defects identified on imaging are not excluded.)
* Contraindication to antiangiogenic agents, including:
* Serious non-healing wound, non-healing ulcer, or bone fracture
* Major surgical procedure or significant traumatic injury within 4 weeks prior to initiating study treatment
* Pulmonary hemorrhage/bleeding event ≥ grade 2 (CTCAE v4.0) within 12 weeks prior to initiating study treatment
* Any other hemorrhage/bleeding event ≥ grade 3 (CTCAE v4.0) within 12 weeks prior to initiating study treatment
* Systolic blood pressure (BP) > 160 mmHg or diastolic BP > 100 mmHg despite optimal medical management
* QT interval, corrected (QTc) > 480 ms (≥ grade 2) on a 12-lead electrocardiogram (ECG)
* If baseline QTc on screening ECG is ≥ grade 2:
* Check potassium and magnesium serum levels
* Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm exclusion of patient due to QTc
* For patients with heart rate < 60 bpm or > 100 bpm, manual read of the QT interval by a cardiologist is required, with Fridericia correction applied to determine QT interval with correction using Fridericia's formula (QTcF) which must be used to determine eligibility (Note: If heart rate is 60-100 bpm, manual read of the QT interval and correction to QTcF is not required).
* Active or clinically significant cardiac disease including any of the following:
* Unstable angina (eg, anginal symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
* Myocardial infarction within 6 months prior to initiating study treatment
* Ventricular arrhythmias requiring anti-arrhythmic therapy other than beta blockers
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Serious (ie, ≥ grade 3) uncontrolled infection
* Uncontrolled effusion
* Known human immunodeficiency virus (HIV) seropositivity (Note: HIV testing is not required)
* Chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Seizure disorder requiring enzyme-inducing anti-epileptic drugs (EIAEDs) (Note: If the seizure disorder can be managed with agents that are not EIAEDs (eg, levetiracetam or valproate), the patient should not be excluded).
* Planned ongoing treatment with other drugs thought to potentially have adverse interactions with either of the study drugs; if such drugs have been used, patients must have discontinued these agents at least 2 weeks (or as noted below) prior to initiating study treatment. Examples include:
* STRONG CYP3A4 inducers

  *Note: Examples of clinical inducers of cytochrome p450 (CYP) isozymes and classification of strong, moderate, and weak interactions are available through the FDA website (Table 3-3 of website:): http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm
* Immunosuppressants (eg, tacrolimus, leflunomide, tofacitinib, roflumilast, pimecrolimus)
* NSAIDs (Note: NSAIDs must be discontinued within 5 days prior to initiating study treatment)
* Pregnancy or breastfeeding
* Previous malignancy with the following exceptions: adequately treated basal cell carcinoma or squamous cell carcinoma of the skin; any in situ malignancy; adequately treated Stage 1 and Stage 2 cancer from which the patient is currently in remission; any other cancer from which the patient has been disease-free for 3 years
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- B: Pemetrexed + Sorafenib: Pemetrexed 375mg/m2 intravenously (IV) Day 1 + Sorafenib 200mg by mouth twice daily on days 1-5, every 21-days of each cycle.
  Experimental Arm B: Pemetrexed: Treatment schedule is administered on day 1 of each 21-day cycle by Intravenous infusion over 10 minutes with a dose of 375 mg/m2. If necessary, the duration of the pemetrexed infusion may be extended to a maximum of 20 minutes.
  Experimental Arm B: Sorafenib: Treatment schedule is administered twice daily by mouth on an empty stomach on days 1-5 of each 21-day cycle with a dose of 200 mg.
Period: Overall Study
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
Started | 9 | 4
Completed | 9 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Continuous [Mean (Full Range); unit: Years] | 54.89 [34 to 65] | 56.75 [43 to 67] | 55.46 [34 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Objective Response Either Partial Response (PR) or Complete Response(CR).
Description: The primary endpoint is the percentage of patients with HER2-negative metastatic breast cancer achieving an objective response (either PR or CR). Overall Response = CR+PR, based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
Time Frame: 2 years 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
Number analyzed (Participants) | 9 | 4
Participants
  Partial Response | 2 | 1
  Stable Disease | 1 | 1
  Progressive Disease | 5 | 0
  Not Evaluable for Response | 1 | 2

2. Secondary Outcome: The Duration of Progression-free Survival (PFS).
Description: Progression-free survival (PFS) defined as the time (in days) from initiation of study treatment until documented disease progression or death, whichever occurs first.
Time Frame: 2 years 3 months
Measure: Number; unit: Days
Groups:
- A: Pemetrexed + Sorafenib: Pemetrexed 500mg/m2 IV Day 1 + Sorafenib 400mg PO BID Days 1-5, Every 14 Days
- B: Pemetrexed + Sorafenib: Pemetrexed 375mg/m2 IV Day 1 + Sorafenib 200mg PO BID Days 1-5, Every 21 Days
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
Number analyzed (Participants) | 9 | 4
Days
  Participant A | 141 | NA — Participant A participated in Arm A only.
  Participant B | 60 | NA — Participant B participated in Arm A only.
  Participant C | 28 | NA — Participant C participated in Arm A only.
  Participant D | 120 | NA — Participant D participated in Arm A only.
  Participant E | 259 | NA — Participant E participated in Arm A only.
  Participant F | 59 | NA — Participant F participated in Arm A only.
  Participant G | 64 | NA — Participant G participated in Arm A only.
  Participant H | 49 | NA — Participant H participated in Arm A only.
  Participant I | 56 | NA — Participant I participated in Arm A only.
  Participant J | NA — Participant J participated in Arm B only. | 22
  Participant K | NA — Participant K participated in Arm B only. | 100
  Participant L | NA — Participant L participated in Arm B only. | 160
  Participant M | NA — Participant M participated in Arm B only. | 19

3. Secondary Outcome: The 2-year Survival Rate After Initial Study Treatment.
Description: The proportion of patients who are alive at 2 years following initiation of study treatment.
Time Frame: 2 years 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
Number analyzed (Participants) | 9 | 4
Participants | 1 | 0

4. Secondary Outcome: Number of Participants at Risk and Affected by Adverse Events (AEs)
Description: To further characterize the safety and side effect profile of the combination. All participants' AEs will be listed and summary descriptive statistics will be calculated.The Adverse events (AEs) are reported using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
Time Frame: 2 years 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
Number analyzed (Participants) | 9 | 4
Participants
  At Risk | 9 | 4
  Affected | 9 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over three years, four months.
Arm/Group | A: Pemetrexed + Sorafenib | B: Pemetrexed + Sorafenib
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/9 | 3/4
Other Adverse Events (participants affected / at risk) | 9/9 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Pemetrexed + Sorafenib (N=9) | B: Pemetrexed + Sorafenib (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Disorders- Other, Specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Gallbladder Obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (3)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Pemetrexed + Sorafenib (N=9) | B: Pemetrexed + Sorafenib (N=4)
Anemia (Blood and lymphatic system disorders) | 9 (15) | 4 (5)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (11) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 7 (10) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (6)
Nausea (Gastrointestinal disorders) | 6 (10) | 4 (8)
Vomiting (Gastrointestinal disorders) | 5 (7) | 3 (4)
Chills (General disorders) | 2 (2) | 2 (3)
Edema limbs (General disorders) | 3 (3) | 1 (2)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (14) | 4 (10)
Fever (General disorders) | 3 (5) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 5 (8) | 4 (6)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 2 (5) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2) | 2 (4)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2)
Alkaline phosphatase increased (Investigations) | 4 (5) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1)
Creatinine increased (Investigations) | 5 (8) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (6) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (9) | 2 (4)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 4 (7) | 2 (2)
Weight loss (Investigations) | 2 (3) | 1 (2)
White blood cell decreased (Investigations) | 4 (6) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 8 (12) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 5 (11) | 4 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (11) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (10) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (8) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (8) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7) | 2 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (6) | 1 (2)
Dysgeusia (Nervous system disorders) | 2 (4) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 3 (5)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (3) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (9) | 1 (4)
Hypotension (Vascular disorders) | 3 (7) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Incomplete objectives due to early termination of trial. Amendment to allow more heavily pretreated subjects to be enrolled required a change in starting doses (Arm B) for all subsequently enrolled subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT02624700/Prot_SAP_000.pdf